CLINICAL TRIAL: NCT04477837
Title: Prospective, Observational, Non-interventional Open-label Multicenter Registry Regarding the Incidence of Heavy Menstrual Bleeding in Women of Reproductive Age Treated With Direct Oral Anticoagulants Because of Venous Thromboembolism
Brief Title: Prospective Comparison of Incidence of Heavy Menstrual Bleeding in Women Treated With Direct Oral Anticoagulants
Status: Completed | Type: Observational
Sponsor: Cardioangiologisches Centrum Bethanien (Other)
Responsible Party: Principal Investigator, Prof. Dr. med. E. Lindhoff-Last, Clinical Professor, Cardioangiologisches Centrum Bethanien
Other Study IDs: HEMBLED
Record Dates: First submitted 2020-07-14; First posted 2020-07-20 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Heavy Menstrual Bleeding
MeSH Terms: conditions — Menorrhagia | interventions — apixaban; Rivaroxaban; edoxaban; Dabigatran

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

GROUPS / COHORTS (4):
- direct oral anticoagulant (DOAC) No.1: Apixaban 5mg, oral, twice daily for at least four months
  Interventions: Drug: Apixaban 5 MG
- direct oral anticoagulant (DOAC) No.2: Rivaroxaban 20mg, oral, once daily for at least four months
  Interventions: Drug: Rivaroxaban 20 MG
- direct oral anticoagulant (DOAC) No.3: Edoxaban 60mg, oral, once daily for at least four months
  Interventions: Drug: Edoxaban 60 MG
- direct oral anticoagulant (DOAC) No.4: Dabigatran 150mg, oral, twice daily for at least four months
  Interventions: Drug: Dabigatran 150 Mg Oral Capsule

INTERVENTIONS:
Drug: Apixaban 5 MG — frequency of heavy menstrual bleeding
  Other Names: Eliquis
  Groups: direct oral anticoagulant (DOAC) No.1
Drug: Rivaroxaban 20 MG — frequency of heavy menstrual bleeding
  Other Names: Xarelto
  Groups: direct oral anticoagulant (DOAC) No.2
Drug: Edoxaban 60 MG — frequency of heavy menstrual bleeding
  Other Names: Lixiana
  Groups: direct oral anticoagulant (DOAC) No.3
Drug: Dabigatran 150 Mg Oral Capsule — frequency of heavy menstrual bleeding
  Other Names: Pradaxa
  Groups: direct oral anticoagulant (DOAC) No.4

SUMMARY:
Prospective comparison of the incidence of heavy menstrual bleeding (HMB) in women of reproductive age treated with direct oral anticoagulants (DOACs)

DETAILED DESCRIPTION:
Patients will be treated as standard of care, no randomization schedule, no blinded investigational product (IP).

The decision which DOAC will be given is made before the subject will enter the trial. The DOAC has to be taken at least for seven days.

The registry is non-interventional (NIS) with routine blood draw at baseline and at month 4 after inclusion. The prospective follow up will be up to four months. Three consecutive menstrual bleeding cycles will be documented by the participating patients at home. One baseline data reporting and one follow up reporting after four months are planned in the participating coagulation centers.

The primary aim is the comparison of the frequency of heavy menstrual bleeding in female patients of reproductive age anticoagulated with DOACs using a modified pictorial blood loss assessment chart.

Secondary aims are the prevalence of von Willebrand disease in young anticoagulated female patients and correlation of HMB with age, International Society of Thrombosis and Hemostasis bleeding assessment tool at inclusion, Blood group, anatomical reasons i.e. underlying uterine pathologies, i. e. presence of uterine fibroids, endometrial polyps and/or adenomyosis, occurrence of iron deficiency, hemoglobin level and intermittent use of non-steroidal anti-inflammatory drug (NSAID).

ELIGIBILITY:
Inclusion Criteria:

* Women with venous thromboembolism
* Age: 18 - 50 years
* Regular menstrual bleeding
* Treatment with DOACs for at least 7 days before inclusion
* Full therapeutic anticoagulation with rivaroxaban 1 x 20 mg, apixaban 2 x 5 mg, edoxaban 60mg once daily or dabigatran 2 x 150mg for at least the next four months
* Written informed consent

Exclusion Criteria:

* Hysterectomy or ovariectomy
* Known heavy menstrual bleeding
* Hormonal contraceptives
* Hormone replacement therapy
* Use of hormone releasing intrauterine System (IUS)
* Contraindications to treatment with DOACs
* Treatment with rivaroxaban 15 mg twice daily (first three weeks after diagnosis of venous thrombosis) or apixaban 10 mg twice daily (first week after diagnosis of venous thrombosis)
* Treatment with rivaroxaban (10 mg or 15 mg once daily) or apixaban (2,5 mg twice daily) in reduced therapeutic dosages
* Participation in any other trial

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Expected number of patients estimated by study duration n=150 patients treated with direct oral anticoagulants (DOAC) due to venous thromboembolism.
Sampling Method: Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-06-15 (Actual)

PRIMARY OUTCOMES:
Primary observation point (for all patients) | baseline and monthly up to month 4
  Frequency of heavy menstrual bleeding in anticoagulated female patients of reproductive Age using a modified Pictorial blood loss assessment Chart (PBAC)-Score (Higham, Br J Obstet Gynaecol 1990; 97: 734-9)

SECONDARY OUTCOMES:
Secondary observation points (for all patients) | up to 16 weeks
  Correlation of heavy menstrual bleeding with von Willebrand's disease; Age; ISTH-BAT-Score at inclusion; blood Group; anatomical reasons i.e. underlying uterine pathologies, i.e. presence of uterine fibroids, endometrial polyps and/or adenomyosis; iron deficiency; hemoglobin level; intermittent use of NSAR

CONTACTS AND LOCATIONS:
Overall Officials: Edelgard Lindhoff-Last, Prof., Principal Investigator — Cardioangiologisches Zentrum Bethanien
Locations (1):
- Cardioangiology Center Bethanien (CCB), Frankfurt am Main, Germany

IPD SHARING:
Plan to Share IPD: No